CLINICAL TRIAL: NCT01384994
Title: Panitumumab After Resection of Liver Metastases From Colorectal Cancer in KRAS Wild-type Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PD Dr. med. Volker Heinemann (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, PD Dr. med. Volker Heinemann, Sponsor Delegatated Person, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PARLIM
Record Dates: First submitted 2011-05-02; First posted 2011-06-29 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Colorectal Cancer; KRAS Wildtype; After Resection of Liver Metastases
Keywords: Colorectal Cancer; PARLIM; KRAS Wildtype; Liver metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folic Acid; Fluorouracil; Oxaliplatin; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FOLFOX + Panitumumab (Experimental)
  Interventions: Drug: Folic Acid; Drug: 5-FU; Drug: Oxaliplatin; Drug: Panitumumab
- FOLFOX (Active Comparator)
  Interventions: Drug: Folic Acid; Drug: 5-FU; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Folic Acid — 400 mg/m2, 2h infusion, d1, q2w
  Arms: FOLFOX + Panitumumab
Drug: 5-FU — 400 mg/m2 bolus iv, d1, q2w
  Arms: FOLFOX + Panitumumab
Drug: 5-FU — 2400 mg/m2 46-h infusion, d1-2, q2w
  Arms: FOLFOX + Panitumumab
Drug: Oxaliplatin — 85 mg/m2 d1, q2w
  Arms: FOLFOX + Panitumumab
Drug: Panitumumab — 6 mg/kg BW every 2 weeks
  Arms: FOLFOX + Panitumumab
Drug: Panitumumab — Panitumumab maintenance phase (3 months) 9mg/kg BW every 3 weeks
  Arms: FOLFOX + Panitumumab
Drug: Folic Acid — 400 mg/m2, 2-h infusion, d1, q2w
  Arms: FOLFOX
Drug: 5-FU — 400 mg/m2 bolus iv, d1, q2w
  Arms: FOLFOX
Drug: 5-FU — 2400 mg/m2 46-h infusion, d1-2, q2w
  Arms: FOLFOX
Drug: Oxaliplatin — 85 mg/m2 d1, q2w
  Arms: FOLFOX

SUMMARY:
Up to 50% of patients with colorectal cancer (CRC) develop liver metastasis during the course of their disease. In 30-40% of patients metastasis is confined to the liver. In these patients R0-resection of metastases may contribute to marked improvement of overall survival. Primary resection of liver metastasis is possible in about 15-20% of patients (Scheele 2005, Petrelli 2005). Recent studies indicate that perioperative chemotherapy may improve survival after resection of liver metastases (Portier 2007, Nordlinger 2007). Nevertheless, there is evidence that 70-80% of patients have recurrent disease after resection of liver metastasis. Stratification for the risk of recurrence may be performed using the FONG-score (Fong 1999).

This study is designed to investigate the efficacy of postoperative chemotherapy combined with an anti-EGFR treatment using panitumumab.

The majority of patients present to the surgeon after chemotherapeutic pretreatment with various not necessarily standardized regimens. Also postoperative therapy after resection of liver metastasis is not a clearly defined standard of care in Germany.

Based on the study by Nordlinger et al. an oxaliplatin-based regimen is chosen for postoperative therapy (Nordlinger 2008). For reasons of practicability mFOLFOX6 was selected as the chemotherapy backbone for additive treatment (Allegra 2010).

Also, there is evidence that the combination of FOLFOX with panitumumab is associated with enhanced antitumor activity (Douillard et al. ESMO 2009). The experimental treatment arm will therefore evaluate the combination of FOLFOX plus panitumumab. Since in colorectal cancer monoclonal antibodies directed against the EGFR are not active in KRAS mutant patients, the experimental arm including panitumumab will only be performed in KRAS wild-type patients (Amado 2008).

The planned study aims to assess the efficacy of postoperative therapy with FOLFOX plus panitumumab followed by maintenance with panitumumab for 3 months in KRAS wild-type patients, compared to the historical data for standard FOLFOX chemotherapy alone, which are verified by a randomised control group without the antibody. (Figure 1: Study Design).

The study will allow preoperative treatment with regimens such as FOLFIRI, XELIRI, FOLFOX or XELOX +/-bevacizumab or +/- cetuximab. However, only those patients will be considered eligible who did not progress during preoperative therapy.

After surgery, a treatment-free interval of at least 4 weeks, but no longer than 8 weeks will be granted.

KRAS-wild-type patients (60% of all pts) will then be randomized in a 2:1 ratio to an experimental arm with FOLFOX + panitumumab or to a reference arm with FOLFOX alone. Combination treatment will be performed for a duration of 3 months, after which patients in the experimental arm will receive maintenance therapy with panitumumab for further 3 months. In the reference arm, treatment will, however, be ended after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided written informed consent.
* R0-resection of liver metastasis, at least four weeks but not longer than 8 weeks ago.
* Histologically confirmed diagnosis of metastatic colorectal cancer confined to the liver
* KRAS-wildtype of the tumor
* Age 18 years or older
* ECOG performance status 0-1
* Females with child-bearing potential must use adequate contraceptive measures
* Exclusion of pregnancy
* Relevant toxicities of previous treatments must have subsided
* Magnesium >= lower limit of normal; Calcium >= lower limit of normal
* Normal cardiac function demonstrated by ECG and echocardiogram (LVEF ≥ 55%)

  * No symptomatic congestive heart failure
  * No unstable angina pectoris
  * No cardiac arrhythmia
* Adequate organ function as defined by Table 1:

  * Hematologic: ANC (absolute neutrophil count) >= 1.5 G/L, Leucocytes > 3.0 G/L, Hemoglobin >= 9 g/dL, Platelets >= 100 G/L
  * Hepatic: Albumin >= 2.5 g/dL, Serum bilirubin <= 2 mg/dL, AST and ALT <= 3 x ULN
  * Renal: Serum Creatinine <= 1.5 mg/dL

Exclusion Criteria:

* Known manifestations of metastatic disease
* Progression during preoperative treatment
* Missing KRAS mutation status of the tumor
* Contraindication against therapy with 5-fluorouracil/ folinic acid or oxaliplatin
* Known intolerability of panitumumab
* Known DPD deficiency
* Polyneuropathy > grade 1 (NCI-CTCv4) which precludes the use of oxaliplatin
* Evidence of ascites or cirrhosis
* Patient is pregnant or lactating or planning to become pregnant within 6 months after end of treatment
* Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment
* Has had a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrolment, or there is an anticipated need for major surgical procedure during the course of the study
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) <= 1 year before enrolment/randomization
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan
* Has a concurrent disease or condition that would make the subject inappropriate for study participation or would interfere with the subject's safety.
* Has any psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Requires concurrent cancer therapy (chemotherapy, radiation therapy, biologic therapy, immunotherapy, or hormonal therapy) while on study.
* Requires concurrent treatment with an investigational agent, participation in another clinical trial, or any specifically prohibited medication while on study.
* Has a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to 5-fluorouracil, folinic acid, oxaliplatin, or panitumumab.
* Other active malignancy
* Known alcohol abuse or drug addiction
* Incapability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years after randomisation

SECONDARY OUTCOMES:
Tolerability and side effects | approximate 6 months after randomisation
Overall Survival | 2 years after randomisation

CONTACTS AND LOCATIONS:
Locations (1):
- Ludwig-Maximilians - University of Munich, Munich, Germany

REFERENCES:
- [Derived] Modest DP, Karthaus M, Kasper S, Moosmann N, Keitel V, Kiani A, Uhlig J, Jacobasch L, Fischer V Weikersthal L, Fuchs M, Kaiser F, Lerchenmuller C, Sent D, Junghanss C, Held S, Lorenzen S, Kaczirek K, Jung A, Stintzing S, Heinemann V. FOLFOX plus panitumumab or FOLFOX alone as additive therapy following R0/1 resection of RAS wild-type colorectal cancer liver metastases - The PARLIM trial (AIO KRK 0314). Eur J Cancer. 2022 Sep;173:297-306. doi: 10.1016/j.ejca.2022.07.012. Epub 2022 Aug 12. PMID 35970102